CLINICAL TRIAL: NCT05327517
Title: Surgery Versus Definitive Chemoradiotherapy for Resectable Cervical Esophageal Squamous Cell Carcinoma: A Prospective Multicenter Open-Label Clinical Trial
Brief Title: Surgery or Chemoradiotherapy for Cervical Esophageal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC3281
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Cervical Esophageal Cancer
Keywords: Esophageal neoplasm; Chemoradiotherapy; Esophagectomy; Overall survival
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Experimental): Patients receive esophagectomy or neoadjuvant therapy plus esophagectomy
  Interventions: Procedure: Esophagectomy
- Definitive chemoradiotherapy (Active Comparator): Patients receive definitive chemoradiotherapy
  Interventions: Procedure: Esophagectomy

INTERVENTIONS:
Procedure: Esophagectomy — Patients receive esophagectomy or definitive chemoradiotherapy according to patient preference
  Other Names: Definitive chemoradiotherapy

SUMMARY:
To compare surgery with definitive chemoradiotherapy for patients with resectable cervical esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resectable cervical esophageal squamous cell carcinoma (cT1b-T4aN0-3M0);
* Cervical esophageal cancers spreads upwards to involve the hypopharynx and downwards to involve the thoracic esophagus can also be included;
* Aged 18-75 years;
* Without any contraindication of operation;
* Hemoglobin >=90 g/L; Leukocytes >=4.0x10^9/L; Absolute neutrophil count >=1.5x10^9/L; Platelet >=100x10^9/L;Total bilirubin <=1.5 ULN; ALT <=2.5 ULN; AST <=2.5 ULN; Serum creatinine <=1.5 ULN or creatinine clearance rate >=50 mL/min (Cocheroft-Gault);INR <=1.5 ULN; APTT <=1.5 ULN;
* Without other malignancies;
* Expected R0 resection;
* ECOG PS 0-1;
* Volunteered to participate in the study, signed the informed consent form.

Exclusion Criteria:

* Without other malignancies;
* With mental diseases;
* With hemorrhagic disease;
* Inoperable patients;
* Pregnant or lactating women;
* Has a history of allergy to paclitaxel or cisplatin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2022-04-10 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 5 years after surgery or definitive Chemoradiotherapy is completed
  5 year overall survival

SECONDARY OUTCOMES:
Laryngo-esophageal dysfunction free survival | 5 years after surgery or definitive Chemoradiotherapy is completed
  5 year laryngo-esophageal dysfunction free survival

CONTACTS AND LOCATIONS:
Overall Officials: Jie He, MD, Study Director — Cancer Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College; Yin Li, MD, Principal Investigator — Cancer Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
expected to be shared as an article paper after the trial ends
Supporting Information: Study Protocol, SAP, CSR
Time Frame: expected to be shared as an article paper after the trial ends